CLINICAL TRIAL: NCT04931082
Title: A Randomized, Double-blinded, Placebo-controlled, Parallel Clinical Trial of a Probiotic on Stress and Cognitive Function in Healthy Adults
Brief Title: Probiotic Intervention for Stress and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Probi AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AFCRO-136
Record Dates: First submitted 2021-06-07; First posted 2021-06-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Stress; Cognition
Keywords: Gut-brain axis; Probiotics
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Active Comparator): One capsule per day for 12 weeks
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): One capsule per day for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — Capsule
  Arms: Probiotics
Dietary Supplement: Placebo — Capsule
  Arms: Placebo

SUMMARY:
The effect of probiotics on stress and cognitive function in healthy adults with moderate stress

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study and comply with its procedures.
* Be able to give written informed consent.
* Be between 21 and 50 years.
* Have moderate stress, as measured on Cohen's Perceived Stress Scale (PSS).
* Are not suffering from depression or anxiety, confirmed by a Hospital Anxiety and Depression Scale (HADS) score.
* Are not regularly consuming probiotics for at least 4 weeks prior to the Screening Visit.
* Is in general good health, as determined by the investigator.

Exclusion Criteria:

* Current diagnosis of currently active irritable bowel syndrome (IBS), according to Rome IV criteria.
* Chronic intestinal disease, immunodeficiency disorder or immunosuppressive treatment.
* Known gluten intolerance, lactose intolerance, milk protein allergy.
* Intake of antibiotics within four weeks prior to the Screening Visit.
* Hypersensitivity to any of the ingredients in the Investigational Product (IP).
* Previous (within 5 years) or ongoing psychiatric illness.
* Consumption of systemic psychotropics, rheumatoid drugs, steroid drugs or creams containing cortisone.
* Regular consumption of asthma medications.
* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk if participating in the study, or influence the results or the participant´s ability to participate in the study.
* Investigator considers the participant unlikely to comply with study procedures, restrictions, and requirements.
* Any disease, that by the investigator's judgement, could interfere with the intestinal barrier function.
* Participation in other clinical trials involving Investigational Product consumption in the last month.
* Desire and/or plans on changing current diet and/or exercise regime during the participation of this trial.
* Participants who are pregnant, breastfeeding, or wish to become pregnant during the study.
* Participants currently of childbearing potential, but not using an effective method of contraception.
* Have a malignant disease or any concomitant end-stage organ disease, which, in the Investigator's judgment, contraindicates participation in the study.
* Individuals who, in the opinion of the investigator, are considered to be poor clinical attendees or unlikely for any reason to be able to comply with the trial.
* Taking any supplements or vitamins notably known to affect cognitive function. Vitamin D and calcium supplements permitted if on a stable dose for the previous 3 months.
* History of heavy caffeinated beverage consumption (>400 mg caffeine/day) within past 2 weeks prior to the Screening Visit.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Determine whether intake of probiotics reduce perceived stress | 12 weeks
  Perceived stress will be evaluated with Cohen's Perceived Stress Scale (PSS) (min 0, max 40)

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantia Food Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No